CLINICAL TRIAL: NCT01056913
Title: Compression Anastomosis: Initial Clinical Experience With the ColonRingTM
Brief Title: NITI CAR27 (ColonRing) Compression Anastomosis in Colorectal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St John of God Hospital, Vienna (Other)
Responsible Party: Principal Investigator, Bernhard Dauser, MD, MD, St John of God Hospital, Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT2
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2013-12

CONDITIONS: Colonic Neoplasms; Rectal Neoplasms; Diverticulitis; Inflammatory Bowel Diseases; Rectal Prolapse
Keywords: anastomotic leakage; bleeding from the anastomotic region; anastomotic stenosis
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Diverticulitis; Inflammatory Bowel Diseases; Rectal Prolapse; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NITI CAR27 (ColonRing) (Other)
  Interventions: Device: Compression Anastomosis Device; Other: follow-up colonoscopy

INTERVENTIONS:
Device: Compression Anastomosis Device — Restoring intestinal continuity using the NITI CAR27 device
  Other Names: ColonRing; BioDynamix Anastomosis
Other: follow-up colonoscopy — endoscopic exploration of anastomosis after complete healing

SUMMARY:
After resection of diseased segments of the large intestine, the continuity of the intestine has to be restored. This can be done by suturing or with so called stapling devices. In addition since 2 centuries compression rings are used to connect the intestine after resection. The NITICAR27 device is a novel compression anastomosis device. The investigators want to prove if this novel device can be compared to commonly used stapling devices concerning anastomotic leakage, bleeding and stenosis.

ELIGIBILITY:
Inclusion Criteria:

* benign and malign lesions of the colon and rectum

Exclusion Criteria:

* advanced peritonitis (putrid, feculent)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Herbst, MD, FRCS, Principal Investigator — St John of God Hospital, Vienna

REFERENCES:
- [Derived] Dauser B, Winkler T, Loncsar G, Herbst F. Compression anastomosis revisited: prospective audit of short- and medium-term outcomes in 62 rectal anastomoses. World J Surg. 2011 Aug;35(8):1925-32. doi: 10.1007/s00268-011-1135-2. PMID 21541799
- See also: About BioDynamix Anastomosis — http://www.nitisurgical.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NITI CAR27 (ColonRing)
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NITI CAR27 (ColonRing)
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 67 [23 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 32

OUTCOME MEASURES:

1. Primary Outcome: Anastomotic Leakage
Time Frame: 4-8 weeks
Measure: Number; unit: participants
Arm/Group | NITI CAR27 (ColonRing)
Number analyzed (Participants) | 62
participants | 0

2. Secondary Outcome: Clinical Relevant Stenosis
Time Frame: six months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | NITI CAR27 (ColonRing)
Serious Adverse Events (participants affected / at risk) | 2/62
Other Adverse Events (participants affected / at risk) | 0/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NITI CAR27 (ColonRing) (N=62)
Anastomotic stenosis (Gastrointestinal disorders) | 2 (2) — Symptomatic anastomotic stenosis resolved by endoscopic dilatation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No